CLINICAL TRIAL: NCT02176122
Title: Randomized Controlled Trial of Meropenem Versus Piperacillin-Tazobactam for Definitive Treatment of Bloodstream Infections Due to Ceftriaxone Non-susceptible E. Coli and Klebsiella Species.
Brief Title: RCT Meropenem vs Piperacillin-Tazobactam for Definitive Treatment of BSI's Due to Ceftriaxone Non-susceptible Escherichia Coli and Klebsiella Spp.
Acronym: MERINO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Secondary to third interim analysis by the study DSMB.
Sponsor: The University of Queensland (Other)
Collaborators: International Society of Chemotherapy (Unknown); Australian Society for Antimicrobials (Unknown); Queensland Clinical Trials & Biostatistics Centre (Unknown); Australasian Society for Infectious Diseases (Other)
Responsible Party: Principal Investigator, Professor David L. Paterson, Professor of Medicine, Infectious Diseases Consultant and Clinical Microbiologist, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTRN12613000532707
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Bloodstream Infections
MeSH Terms: conditions — Sepsis | interventions — Meropenem; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meropenem (Active Comparator): Meropenem 1g adm every 8 hours IV up to study day 4.
  Interventions: Drug: Meropenem
- Piperacillin-tazobactam combination product (Experimental): Piperacillin/tazobactam 4.5g adm every 6 hours IV up to study day 4.
  Interventions: Drug: Piperacillin-tazobactam combination product

INTERVENTIONS:
Drug: Meropenem — Meropenem is a carbapenem anti-bacterial used for the treatment of serious infections in patients.
  Other Names: Merrem; Meronem
  Arms: Meropenem
Drug: Piperacillin-tazobactam combination product — Piperacillin-tazobactam is used for the treatment of patients with systemic and/or local bacterial infections.
  Other Names: Zosyn; Tazocin
  Arms: Piperacillin-tazobactam combination product

SUMMARY:
No randomized controlled trials (RCTs) have yet been performed comparing different treatment options for AmpC or ESBL-producing Enterobacteriaceae. During the last 10 years we have seen an exponentially increasing rate of carbapenem resistance worldwide, including Australia and New Zealand. The investigators urgently need data from well-designed RCTs to guide clinicians in the treatment of antibiotic resistant Gram-negative infections. The investigators face a situation where a commonly used antibiotic for these infections (meropenem) may be driving carbapenem resistance. For this reason, the investigators are seeking to compare a carbapenem-sparing regimen with a carbapenem for the treatment of these infections. Formal evaluation of safety and efficacy of generic antibiotics in the treatment of infection is of immense clinical and public health importance, and no formal trial has yet been conducted to address these issues. The international collaboration between teams of clinician researchers, some of whom are leaders in their field, makes it highly likely that the outcomes of this trial will have a significant impact on clinical practice.

The investigators' hypothesis is that piperacillin/tazobactam (a carbapenem-sparing regimen) is non-inferior to meropenem (a widely used carbapenem) for the definitive treatment of bloodstream infections due to third-generation cephalosporin non-susceptible E. coli or Klebsiella species.

DETAILED DESCRIPTION:
Escherichia coli and Klebsiella spp. are common causes of bacteraemia, and may acquire genes encoding extended-spectrum beta-lactamases (ESBLs) or AmpC beta-lactamases (1). ESBL or AmpC producers are typically resistant to third generation cephalosporins such as ceftriaxone, but susceptible to carbapenems (1). Observational studies have been performed evaluating antibiotic choices for ESBL producers (2-9). In no study has the outcome of treatment for serious infections for ESBL producers been significantly surpassed by carbapenems (2-9).

Despite the potential advantages of carbapenems for treatment of ceftriaxone non-susceptible organisms, widespread use of carbapenems may cause selection pressure leading to carbapenem-resistant organisms. This is a significant issue since carbapenem-resistant organisms are treated with "last-line" antibiotics such as colistin. Some new beta-lactam antibiotics and beta-lactamase inhibitors, which are active against ESBL, AmpC and some carbapenemase producing organisms, are in advanced clinical development (10). However, these antibiotics are likely to be expensive and may best be held in reserve for infections where there are no alternatives. Therefore, we see a need for establishing the efficacy of a generically available alternative to carbapenems for serious infections.

The susceptibility of ESBL producers and AmpC producers to piperacillin/tazobactam is less predictable than that of carbapenems. By definition, ESBLs are inhibited by beta-lactamase inhibitors such as tazobactam (1). However, E. coli or Klebsiella may produce multiple beta-lactamase types some of which are resistant to inhibition by tazobactam. Additionally, in some cases outer membrane protein loss may contribute to resistance to tazobactam. By definition, AmpC is not inhibited by beta-lactamase inhibitors such as tazobactam. However, despite these limitations, approximately 50% or more of ceftriaxone non-susceptible E. coli or Klebsiellae remain susceptible in vitro to piperacillin/tazobactam (1).

No randomised controlled trials have yet been performed comparing different treatment options for ceftriaxone resistant Enterobacteriaceae. The largest observational study with an analysis by treatment outcome was published in February 2012 by Rodriguez-Bano and colleagues (9). They performed a post-hoc analysis of six published cohorts of patients with bacteraemia due to ESBL producing E. coli. Two nonmutually exclusive cohorts (empirical therapy and definitive therapy) were constructed and analysed separately. In both cohorts, carbapenems were not superior to beta-lactam/beta-lactamase inhibitor combinations (BLBLIC). Specifically, in the definitive therapy cohort, mortality rates at 30 days were not significantly different - 9.3% for those who received a BLBLIC and 16.7% for those who received a carbapenem (p>0.20) (9).

ELIGIBILITY:
Inclusion Criteria:

* Bloodstream infection with E. coli or Klebsiella spp. with proven non-susceptibility to third generation cephalosporins and susceptibility to meropenem and piperacillin-tazobactam from at least one blood culture draw. This will be determined in accordance with laboratory methods and susceptibility breakpoints defined by EUCAST standards (www. eucast.org). Bacterial identification to species level will be performed using standard laboratory methods (e.g. MALDI-TOF) and susceptibility testing (e.g. Vitek2)
* No more than 72 hours has elapsed since the first positive blood culture collection.
* Patient is aged 18 years and over
* The patient or approved proxy is able to provide informed consent.

Exclusion Criteria:

* Patient not expected to survive more than 4 days
* Patient allergic to a penicillin or a carbapenem
* Patient with significant polymicrobial bacteraemia (that is, a Gram positive skin contaminant in one set of blood cultures is not regarded as significant polymicrobial bacteraemia).
* Treatment is not with the intent to cure the infection (that is, palliative care is an exclusion).
* Pregnancy or breast-feeding.
* Use of concomitant antimicrobials in the first 4 days after enrolment with known activity against Gram-negative bacilli (except trimethoprim/sulfamethoxazole may be continued as Pneumocystis prophylaxis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2014-02; Primary Completion 2017-07-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Mortality at 30 days | 30 days
  To compare the 30-day mortality post bloodstream infection of piperacillin/tazobactam and meropenem.

SECONDARY OUTCOMES:
Time to clinical and microbiologic resolution of infection | on or before study day 4
  defined as number of days from randomisation to resolution of fever (temperature > 38.0o C) and leucocytosis (white blood cell count >12x109/L) PLUS sterilisation of blood cultures.
Clinical and microbiologic success | day 4
  defined as survival PLUS resolution of fever and leucocytosis PLUS sterilisation of blood cultures
Microbiologic resolution of infection | day 4
  defined as sterility of blood cultures collected on or before day 4
Microbiologic relapse | day 30
  defined as growth of a meropenem resistant Gram negative bacillus from any clinical specimen collected or a positive stool test (according to local lab diagnostic procedures) for C. difficile, from day 4 of study drug administration to day 30
Superinfection with a carbapenem or piperacillin-tazobactam resistant organism or Clostridium Difficile | day 30
  To compare the risk of superinfection with a carbapenem resistant organism with each regimen.

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, PhD, Principal Investigator — UQCCR, RBWH
Locations (31):
- Australia (14):
  - Shellharbour Hospital (Illawarra Shoalhaven Local Health District), Shellharbour, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Brisbane Private Hospital, Brisbane, Queensland
  - St. Andrew's War Memorial Hospital, Brisbane, Queensland
  - Mater Misericordiae Health Services Brisbane Ltd., Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Barwon Health, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth
- Sunnybrook Research Institute, Toronto, Canada
- Italy (6):
  - Teaching Hospital - Sant'Orsola Malpighi, Bologna
  - Dipartimento di Scienze Biomediche e Cliniche "L. Sacco". Azienda Ospedaliera - Polo Universitario, Milan
  - "Sapienza" University of Rome, Rome
  - Catholic University Rome, Rome
  - Sanremo Hospital, Sanremo
  - Santa Maria Misericorida University Hospital, Udine
- The American University of Beirut, Beirut, Lebanon
- New Zealand (2):
  - Middlemore Hospital, Papatoetoe
  - The North Shore Hospital, Westlake
- Saudi Arabia (2):
  - King Fahad Specialist Hospital, Dammam
  - King Saud Bin Abdulaziz University for Health Sciences, King Abdulaziz Medical City, Riyadh
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Africa (2):
  - Groote Schuur Hospital, Cape Town
  - Charlotte Maxeke Johannesberg Academic Hospital, Johannesburg
- İstanbul Medipol Üniversitesi Medipol Mega Hastaneler Kompleksi (Medipol Mega Hospitals Complex), Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Harris PNA, Tambyah PA, Lye DC, Mo Y, Lee TH, Yilmaz M, Alenazi TH, Arabi Y, Falcone M, Bassetti M, Righi E, Rogers BA, Kanj S, Bhally H, Iredell J, Mendelson M, Boyles TH, Looke D, Miyakis S, Walls G, Al Khamis M, Zikri A, Crowe A, Ingram P, Daneman N, Griffin P, Athan E, Lorenc P, Baker P, Roberts L, Beatson SA, Peleg AY, Harris-Brown T, Paterson DL; MERINO Trial Investigators and the Australasian Society for Infectious Disease Clinical Research Network (ASID-CRN). Effect of Piperacillin-Tazobactam vs Meropenem on 30-Day Mortality for Patients With E coli or Klebsiella pneumoniae Bloodstream Infection and Ceftriaxone Resistance: A Randomized Clinical Trial. JAMA. 2018 Sep 11;320(10):984-994. doi: 10.1001/jama.2018.12163. PMID 30208454
- [Derived] Harris PN, Peleg AY, Iredell J, Ingram PR, Miyakis S, Stewardson AJ, Rogers BA, McBryde ES, Roberts JA, Lipman J, Athan E, Paul SK, Baker P, Harris-Brown T, Paterson DL. Meropenem versus piperacillin-tazobactam for definitive treatment of bloodstream infections due to ceftriaxone non-susceptible Escherichia coli and Klebsiella spp (the MERINO trial): study protocol for a randomised controlled trial. Trials. 2015 Jan 27;16:24. doi: 10.1186/s13063-014-0541-9. PMID 25623485